CLINICAL TRIAL: NCT04628819
Title: Effect and Tolerability of Lactobacillus Rhamnosus GG LA801 for the Preventive Nutritional Care of Nosocomial Diarrhea in Children
Acronym: EPISODE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Not enough patients included
Sponsor: PiLeJe (Industry)
Collaborators: Clinact (Other); Clinfile (Industry)
Responsible Party: Sponsor
Organization: Larena SAS (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2019-A01797-50; 2019-A01797-50 (Other: ANSM (ID-RCB)); 19.07.30.37834 (Other: CNRIPH (French Ethic Committee))
Record Dates: First submitted 2020-11-09; First posted 2020-11-16 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Nosocomial Infection; Diarrhea, Infantile
Keywords: Lactobacillus Rhamnosus; Children; Dietary Supplementation; Preventive nutritional care
MeSH Terms: conditions — Cross Infection; Diarrhea, Infantile

STUDY DESIGN:
Intervention Model Description: Patients will be randomized in one of the two parallel groups. The first group will be supplemented with Lactobacillus Rhamnosus and the second group will intake a placebo.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The patients, their parents and the investigators will not know the treatment taken by the patient. Unblinding will be performed at the end of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Babybiane Imedia (Experimental): Patients receive Babybiane Imedia once daily during seven days.
  Interventions: Dietary Supplement: Babybiane Imedia or placebo
- Placebo (Placebo Comparator): Patients receive a placebo with the same consistency and taste as the Babybiane Imedia once daily during seven days.
  Interventions: Dietary Supplement: Babybiane Imedia or placebo

INTERVENTIONS:
Dietary Supplement: Babybiane Imedia or placebo — Both the investigational product as well as the placebo will be administered once daily, diluted in a nursing bottle or a glass of water or cold milk, or mixed with a food suitable for the child. It may be diluted in oral rehydration solution and is to be taken preferably before a meal. Both preparations (BABYBIANE® Imedia and placebo) will have similar consistency and taste. A supplementation unit will contain 7 packs of either products, one per supplementation day.

SUMMARY:
One of the most common infections acquired in hospital, also known as nosocomial infections, is intestinal infections. These infections can lead to the development of nosocomial diarrhea which can have serious consequences in young / very young children. These infections tend to prolong the average length of hospital stay of this fragile population. Conventional treatment of these infections, in the absence of knowledge of the infectious agent, is purely symptomatic. It is therefore necessary to develop new prevention strategies for this type of disease. In this sense, the administration of probiotic strains in order to prevent the onset of nosocomial diarrhea is a promising avenue and the present study aims to validate the preventive effect of this supplement.

The objective of this study is to assess the effect of Babybiane® Imedia or the microbiotic strain Lactobacillus rhamnosus GG LA801 in the preventive nutritional management of nosocomial diarrhea in children aged 1 to 24 months. This evaluation will be made in comparison with a placebo. The tolerance of the product under study will also be assessed.

DETAILED DESCRIPTION:
Diarrhea in children According to the World Health Organization, diarrhea is defined by the release of at least three loose or watery stools per day or with an abnormal frequency for a single individual. It is generally a symptom of gastrointestinal infection who might be of bacterial or viral, parasite origin. Acute diarrhea is a frequent pathology, with an infectious origin in most of the cases, especially viruses and bacteria in industrialized countries. It leads to a risk of acute dehydration, in particular in high-risk populations as newborns, infants and toddlers.

Acute diarrhea is still the second leading cause of infection-associated death of children under five worldwide and in 2011 it was estimated to account for almost 10 % of the 7 million deaths in that population. In European countries, most cases show only mild or moderate symptoms and fatal outcomes are very uncommon. However gastroenteritis is still one of the main reasons for hospitalization of children in this region. In Europe, the incidence or diarrhea ranges from 0.5 to 2 episodes per year in children under 3 years old. Dehydration secondary to an acute diarrhea is still one of the main cause of death in young children that could be prevented in industrialized countries. Acute diarrhea is mostly associated with acute gastroenteritis, which is one of the main reason for hospitalization of children under 3 but it is also associated with antibiotics therapy (Antibiotics Associated Diarrhea or AAD) or hospital-acquired infections.

Hospital-acquired or nosocomial diarrhea (ND) Infections occurring more than 48 hours after hospital admission are usually considered as nosocomial infections. The incidence of this kind of infections among children in the industrialized countries remains very high, ranging from 5.1% to 11.6% depending on the time of the year and the type of hospital. In children, gastrointestinal infections account for the majority of the hospital-acquired infections and rotavirus is the main pathogenic agent. Those infections can lead to nosocomial diarrhea and therefore have numerous health and economic consequences as they tend to prolong hospital stay and mortality. Moreover nosocomial infections are usually treated with broad spectrum antibiotics without knowing the type of bacteria responsible for the infection or its antibiogram. This results in the selection of resistant microorganisms leading to increased antimicrobial resistance. All these factors combine for an increase of the financial burden of the healthcare system due to nosocomial infections. Nosocomial infections are more prevalent in the pediatric population than in the adult population and predominantly occur in intensive care units (ICU). In settings other than the ICU, the most common pediatric nosocomial infection is gastroenteritis. Rotavirus and norovirus account for the vast majority of the hospital-acquired gastroenteritis. Although, regular precautions such as hand hygiene or isolation of sick patients can prevent the spread of the infections, there is a clear need for new prevention strategies, and among those the use of probiotics is a promising one.

Probiotics and nosocomial diarrhea It is important to consider that no broad consensus exists to recommend the use of probiotics in the prevention of diarrhea, mainly because of the different design of the studies done so far. Therefore, there is a need for more well-designed studies before recommendations can be proposed.

However, three systematic reviews have assessed the efficacy of probiotics supplementation in the prevention of nosocomial diarrhea for a total of eight randomized clinical trials (RCT) involving a grand total of 2 254 children for the age of 1 month to 18 years old.

The characteristics and results of these RCTs are summarized in the following tables:

The analysis of the results of these clinical trials revealed that among all the probiotics strains tested, only Lactobacillus rhamnosus GG (LGG) was proved to be efficient in reducing the risk for nosocomial rotavirus-associated diarrhea. Differential effects have been observed depending on the intestinal pathogen, thus it would be interesting to analyze the pathogenic agent responsible for the diarrhea observed in the study participants.

Based on the aforementioned meta-analysis, and although it is not a formal recommendation, the European Society for Paediatric Gastroenterology Hepatology and Nutrition (ESPGHAN) working group strongly suggests the use of Lactobacillus rhamnosus GG (≥109 CFU/day over the course of the hospital stay) to prevent nosocomial diarrhea in children. It is important to consider that LGG is the only probiotic strain for which available data were deemed sufficient to lead to a recommendation.

Mechanism of action of Lactobacillus rhamnosus GG Multiple studies have shown that Lactobacilli increase mucin secretion by intestinal epithelial cell lines in vitro, increase tight junction protein expression, thus preventing damaging action from pathogenic bacteria. Probiotics such as lactobacillus spp. can also exert an antimicrobial activity by producing short chain fatty acids. In addition, probiotics can inhibit virus adsorption by competing with viral receptors on intestinal cells and can also have a beneficial effect on parasitic infections.

Moreover, several studies have previously shown that LGG increases mucosal secretory immunoglobulin A and inhibits viral adhesion on intestinal epithelial cell surface, inhibits virion secretion, and reduces viral replication in the mucosa. LGG also enhances immune response targeted against rotavirus by stimulating rotavirus-specific interferon (IFN)-γ-production from T-Cells. In addition, LGG reduces the rotavirus-induced release of reactive oxygen species in vitro and suppresses the rotavirus-induced interleukin (IL)-6 response in a non-transformed porcine intestinal epithelial cell line. Finally LGG has been shown to increase Nitric oxide production in epithelial intestinal cells in vitro, hence increasing antimicrobial activity.

In conclusion, in light of all the available data on the potential beneficial effect of LGG on intestinal infections, dietary supplementation with Lactobacillus rhamnosus GG to a dose of ≥1.1010 CFU/day and in addition to an oral rehydration solution, in line with the recommendations of the international institutions (American Academy of Pediatrics, ESPGHAN, European Society for Paediatric Infectious Diseases, GFHGNP, World Gastroenterology Organization) in regards to the nutritional care of acute diarrhea in children seems promising.

The present study is designed to assess the effect of Laboratoires PiLeJe own Lactobacillus rhamnosus GG LA801 formula in reducing the incidence of nosocomial diarrhea in children under 24 months who stayed in an emergency department for whatever medical reason and for over 6 hours.

Product indications and contra-indications BABYBIANE® Imedia is a food for special medical purposes containing Lactobacillus rhamnosus intended for nutritional care of newborns and young children suffering from acute diarrhea.

From a regulatory standpoint, this product is within the following context:

* Regulation (UE) No 609/2013 of the European parliament and of the 12/06/2013 council related to the dietary products destined for newborns and infants, food for special medical purposes and substitutes of the total daily intake for weight control;
* Regulation (EU) 2016/128 supplementing Regulation (EU) No 609/2013 of the European Parliament and of the Council as regards the specific compositional and information requirements for food for special medical purposes.

Regulation (UE) No 609/2013 does not significantly modify the former definition of a food for special medical purposes (FSMP) defined as being a "dietary product specifically treated and formulated and destined to satisfy dietary needs of patients, including newborns, and that can only be used under medical supervision and destined to be the exclusive or partial diet of the patients whose capabilities of absorption, digestion, assimilation, metabolization or excretion of regular food products or some of their ingredients or metabolites are diminished, limited or altered or whose health status determine other specific dietary demands that cannot be satisfied only by a modification of the regular diet".

FSMPs are ranked into three different categories. BABYBIANE® Imedia falls into the third category: "nutritionally incomplete food product, whose composition is adapted to fulfill the specific needs of newborns and young children with acute diarrhea and which cannot be the only food source."

Indications BABYBIANE® Imedia contains ≥1.1010 Colony Forming Units (CFU) of Lactobacillus rhamnosus GG LA801 per pack and is strongly recommended for nutritional care of acute diarrhea (associated with acute gastro enteritis, antibiotics therapy or hospital-acquired) in newborns or young children.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent signed by the patient's legal guardian(s) for study enrollment;
* Aged 1 to 24 months ;
* Admitted to the hospital for reasons other than diarrhea;
* Stayed in the Short Stay Unit, SSU, for a minimum duration of 6h.

Exclusion Criteria

* With history of gastroenteritis in the 2 weeks before hospitalization;
* With symptoms suggesting an ongoing gastroenteritis or other intestinal disease;
* Use of probiotics or prebiotics within 7 days before admission;
* With immunodeficiency, neoplasm or chronic severe illnesses;
* With a previous hospitalization within 15 days;
* With an history of digestive surgery;
* For whom an oral route is impossible;
* Participating at the same time in another clinical trial.

Ages: 1 Month to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 61 (Actual)
Dates: Start 2019-12-29 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
incidence of nosocomial diarrhea | during seven days of supplementation
  The primary endpoint is the comparison of the incidence of nosocomial diarrhea (defined as the passage of 3 or more loose or watery stools in a 24-hour period (or more frequently than is normal for the individual) that occurred between 48 hours to 7 days after admission) between the 2 groups (BABYBIANE® Imedia vs. placebo) during 7 days of supplementation.

SECONDARY OUTCOMES:
time to onset of nosocomial diarrhea | During study duration (14 days)
  Comparison of time to onset of nosocomial diarrhea between the 2 groups
number of nosocomial diarrhea | During study duration (14 days)
  Comparison of the number of nosocomial diarrhea between the 2 groups
nosocomial diarrhea duration | During study duration (14 days)
  Comparison of nosocomial diarrhea duration (defined as the time until the last loose watery stools from the onset of diarrhea that occurs between 48 hours to 7 days after admission) between the 2 groups
incidence of diarrhea | During study duration (14 days)
  Comparison of incidence of diarrhea (defined as the passage of 3 or more loose or watery stools in a 24-hour period (or more frequently than is normal for the individual)) between the 2 groups for the whole duration of a patient's study participation (i.e. 14 days)
time to onset of diarrhea | During study duration (14 days)
  Comparison of time to onset of diarrhea between the 2 groups
number of loose or watery stools | During study duration (14 days)
  Comparison of the number of loose or watery stools between the 2 groups
diarrhea duration | During study duration (14 days)
  Comparison of diarrhea duration (defined as the time until the last loose watery stools from the onset of diarrhea) between the 2 groups
incidence of recurrent diarrhea | During study duration (14 days)
  Comparison of incidence of recurrent diarrhea (after 48 hours of normal stools) between the 2 groups
incidence of need for and length of rehydration because of diarrhea | During study duration (14 days)
  Comparison of incidence of need for and length of rehydration because of diarrhea between the 2 groups
length of hospital stay | During study duration (14 days)
  Comparison of length of hospital stay between the 2 groups
number of care visits | During study duration (14 days)
  Comparison of number of care visits between the 2 groups
length of day care missed | During study duration (14 days)
  Comparison of length of day care missed between the 2 groups
length of work missed by parent or guardian | During study duration (14 days)
  Comparison of length of work missed by parent or guardian between the 2 groups
other symptoms presence | During study duration (14 days)
  Comparison of other symptoms presence between the 2 groups : fever, vomiting, respiratory infections, etc
rotavirus, viral or bacterial pathogens' presence on stools | During study duration (14 days)
  Comparison of rotavirus, viral or bacterial pathogens' presence on stools between the 2 groups
adverse events | During study duration (14 days)
  Comparison of adverse events (rate of patients, type of events, relation with the complementation …) between the 2 groups
Complementation intake | During study duration (14 days)
  Comparison of observance (percentage of diluted complementation consumed per day) between the 2 groups

CONTACTS AND LOCATIONS:
Overall Officials: Alexis Mosca, MD, Principal Investigator — Hopital Universitaire Robert-Debre
Locations (2):
- France (2):
  - Centre hospitalier d'Auxerre, Auxerre
  - Hopital Robert Debré, Paris

IPD SHARING:
Plan to Share IPD: No